CLINICAL TRIAL: NCT05241236
Title: Office Based MRI/Ultrasound Guided Prostate Cancer Ablation: Outcomes Registry
Brief Title: MRI/Ultrasound Fusion Guided Laser Ablation of Prostate Cancer
Acronym: MRFLA
Status: Recruiting | Type: Observational
Sponsor: Urological Research Network, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: URN-20-014
Record Dates: First submitted 2021-09-26; First posted 2022-02-15 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Neoplasms Prostate; Cancer of the Prostate
Keywords: Prostate; PSA; FUSION; Ultrasound; MRI; Cancer; Laser; Outcomes; Recurrence; QOL, Quality of Life; Urinary function; Sexual Function
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Image Fusion (MR/US) Software Registration Guided Laser Ablation of Prostate Cancer — Subjects diagnosed by a transperineal fusion or random transperineal or random transrectal prostate biopsy. Laser treatment plan generated by biopsy results +/- MRI is uploaded into the device. In procedure suite, a transperineal anesthetic block is conducted following by Bianco - USPTO PCT/US18/24404. On lithotomy a transrectal ultrasound probe is advanced, the prostate scanned. The images are acquired by fusion device. Co-registration is performed by surgeon delimiting boundaries of prostate. Medical device delivers real-time fusion guidance outlining prostate contours, ablation goals and laser introduce location. Surgeon executes plan or adjust as needed. Surgeon activates laser device, performs ablation monitored by medical device in real-time. The fusion device will deliver great perspective between the ablation areas and critical anatomical landmarks such as: NVB, membranous urethra, etc. Patient is dismissed to the recovery room and discharged afterwards
  Other Names: Intervention of Interest: Prostate Cancer Laser Ablation

SUMMARY:
This serves as a registration trial. It aims to record short, intermediate, and long-term outcomes of patients treated with targeted laser ablation of biopsy confirmed prostate cancer. Outcomes will be categorized as: 1- Procedure Related, 2- Perioperative - Adverse Events that may occur within 90 days, 3-Oncologic: Recurrence of cancer in treatment area, de-novo tumors, conversion to radical surgery, radiation or cryoablation, emergence of metastasis, 4- Functional: Sexual and Urinary function following treatment

DETAILED DESCRIPTION:
CLINICAL REGISTRY OBSERVATION NATURE

This serves as a registration trial evaluating short, intermediate, and long-term outcomes of patients treated with targeted laser ablation of biopsy confirmed prostate cancer. The primary outcome measure is 1-year oncological control of the targeted ablated area. The following secondary aims are sought: PROCEDURE RELATED: tolerability, feasibility, pain during this office-based procedure. PERIOPERATIVE: Adverse Events (AEs) and Series AEs profile during the initial 90 days after the procedure. ONCOLOGIC - In addition to primary aim, determine risk and rate of emergence of de-novo tumors (so called Outfield Recurrence) at the 1 year fusion biopsy mark and overtime. Will also observe rate of progression locally and systemically. Conversion to whole gland treatment - surgery extraction, radiation or whole gland cryoablation is of particular interest as is the initiation of androgen suppression (castration). Moreover, the investigators will evaluate the impact of MRI in assessing tumor locations and of software registration guiding the location and extent of ablation of the laser ablation over fixed time intervals. Finally, incidence of metastatic disease - non castrate and castrate - as well as cancer specific and overall survival at 5, 10 and 15 years post procedure. FUNCTIONAL OUTCOMES - determine urinary function and sexual function including incidence of ejaculation, and climacturia at months 3, 6 and 12. These outcomes will then measured yearly for the extent of the study

ELIGIBILITY:
Inclusion Criteria:

* Men between 50 and 65 years of age with a clinical diagnosis of prostate cancer with Low or Intermediate risk prostate cancer, and <50% positive core rate by prostate lobe
* Men older than 65 years of age with clinical diagnosis of prostate cancer <50% positive core rate by prostate lobe
* Absence of extra-capsular extension
* Absence of seminal vesicle invasion
* Absence of regional or distant metastatic disease
* Multiparametric MRI of the prostate performed either before the biopsy or >10 weeks after prostate biopsy
* Treated with Cryotherapy of the prostate
* Treatment based on co-registration between MP-MRI and Prostate Ultrasound

Exclusion Criteria:

* Prior treatment of prostate cancer in the form of surgery.
* Performance status greater than 0 based on ECOG criteria
* Mental status impairment

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As written in Initial Section
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2038-11 (Estimated)

PRIMARY OUTCOMES:
Primary Oncological Control | 1 Year
  Negative CANCER Rate in treated area after fusion biopsy

SECONDARY OUTCOMES:
Perioperative Outcomes | 90 days
  Rate of Adverse Events and Serious Adverse Events following CTCAE v5 classification
Urinary Function | 5 years
  Rate of AUA symptoms score less than 7 (Scale 0-35).
Sexual Function | 5 years
  Rate of Sexual Inventory for men scores above 15 (Scale 1-25)
Radiological Cancer Control | 5 Years
  Rate of Detection of discrete lesions following multi-parametric prostate MRI

OTHER OUTCOMES:
Rate of Conversion to Whole gland treatment - Salvage Treatment | 10 years
  Conversion to radical surgery or radiation or cryoablation
Rate of development of metastasis | 10 years
  Detection of metastatic disease

CONTACTS AND LOCATIONS:
Overall Officials: FERNANDO J BIANCO, MD, Principal Investigator — UROLOGICAL RESEARCH NETWORK; EUSEBIO LUNA, MD, Study Director — UROLOGICAL RESEARCH NETWORK; Isabel H Lopez, MD, Study Director — UROLOGICAL RESEARCH NETWORK
Locations (1):
- Urological Research Network, Miami Lakes, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Non identifiable pertinent information will be shared for other scientists to evaluate other pertinent questions
Supporting Information: CSR
Time Frame: 6 years
Access Criteria: institutional agreement, HIPPA compliance

REFERENCES:
- [Background] Moore CM, Kasivisvanathan V, Eggener S, Emberton M, Futterer JJ, Gill IS, Grubb Iii RL, Hadaschik B, Klotz L, Margolis DJ, Marks LS, Melamed J, Oto A, Palmer SL, Pinto P, Puech P, Punwani S, Rosenkrantz AB, Schoots IG, Simon R, Taneja SS, Turkbey B, Ukimura O, van der Meulen J, Villers A, Watanabe Y; START Consortium. Standards of reporting for MRI-targeted biopsy studies (START) of the prostate: recommendations from an International Working Group. Eur Urol. 2013 Oct;64(4):544-52. doi: 10.1016/j.eururo.2013.03.030. Epub 2013 Mar 20. PMID 23537686
- [Background] Costa DN, Pedrosa I, Donato F Jr, Roehrborn CG, Rofsky NM. MR Imaging-Transrectal US Fusion for Targeted Prostate Biopsies: Implications for Diagnosis and Clinical Management. Radiographics. 2015 May-Jun;35(3):696-708. doi: 10.1148/rg.2015140058. Epub 2015 Mar 18. PMID 25786055
- [Background] Barentsz JO, Richenberg J, Clements R, Choyke P, Verma S, Villeirs G, Rouviere O, Logager V, Futterer JJ; European Society of Urogenital Radiology. ESUR prostate MR guidelines 2012. Eur Radiol. 2012 Apr;22(4):746-57. doi: 10.1007/s00330-011-2377-y. Epub 2012 Feb 10. PMID 22322308
- [Background] Eldred-Evans D, Neves JB, Simmons LAM, Kanthabalan A, McCartan N, Shah TT, Arya M, Charman SC, Freeman A, Moore CM, Punwani S, Emberton M, Ahmed HU. Added value of diffusion-weighted images and dynamic contrast enhancement in multiparametric magnetic resonance imaging for the detection of clinically significant prostate cancer in the PICTURE trial. BJU Int. 2020 Mar;125(3):391-398. doi: 10.1111/bju.14953. Epub 2019 Dec 11. PMID 31733173
- [Background] Simmons LAM, Kanthabalan A, Arya M, Briggs T, Barratt D, Charman SC, Freeman A, Hawkes D, Hu Y, Jameson C, McCartan N, Moore CM, Punwani S, van der Muelen J, Emberton M, Ahmed HU. Accuracy of Transperineal Targeted Prostate Biopsies, Visual Estimation and Image Fusion in Men Needing Repeat Biopsy in the PICTURE Trial. J Urol. 2018 Dec;200(6):1227-1234. doi: 10.1016/j.juro.2018.07.001. Epub 2018 Jul 11. PMID 30017964
- [Background] Hamid S, Donaldson IA, Hu Y, Rodell R, Villarini B, Bonmati E, Tranter P, Punwani S, Sidhu HS, Willis S, van der Meulen J, Hawkes D, McCartan N, Potyka I, Williams NR, Brew-Graves C, Freeman A, Moore CM, Barratt D, Emberton M, Ahmed HU. The SmartTarget Biopsy Trial: A Prospective, Within-person Randomised, Blinded Trial Comparing the Accuracy of Visual-registration and Magnetic Resonance Imaging/Ultrasound Image-fusion Targeted Biopsies for Prostate Cancer Risk Stratification. Eur Urol. 2019 May;75(5):733-740. doi: 10.1016/j.eururo.2018.08.007. Epub 2018 Dec 6. PMID 30527787
- [Background] Bonmati E, Hu Y, Villarini B, Rodell R, Martin P, Han L, Donaldson I, Ahmed HU, Moore CM, Emberton M, Barratt DC. Technical Note: Error metrics for estimating the accuracy of needle/instrument placement during transperineal magnetic resonance/ultrasound-guided prostate interventions. Med Phys. 2018 Apr;45(4):1408-1414. doi: 10.1002/mp.12814. Epub 2018 Mar 9. PMID 29443386
- [Background] Orczyk C, Barratt D, Brew-Graves C, Peng Hu Y, Freeman A, McCartan N, Potyka I, Ramachandran N, Rodell R, Williams NR, Emberton M, Ahmed HU. Prostate Radiofrequency Focal Ablation (ProRAFT) Trial: A Prospective Development Study Evaluating a Bipolar Radiofrequency Device to Treat Prostate Cancer. J Urol. 2021 Apr;205(4):1090-1099. doi: 10.1097/JU.0000000000001567. Epub 2020 Dec 14. PMID 33315505
- [Background] Simmons LAM, Kanthabalan A, Arya M, Briggs T, Barratt D, Charman SC, Freeman A, Gelister J, Hawkes D, Hu Y, Jameson C, McCartan N, Moore CM, Punwani S, Ramachandran N, van der Meulen J, Emberton M, Ahmed HU. The PICTURE study: diagnostic accuracy of multiparametric MRI in men requiring a repeat prostate biopsy. Br J Cancer. 2017 Apr 25;116(9):1159-1165. doi: 10.1038/bjc.2017.57. Epub 2017 Mar 28. PMID 28350785
- [Background] Bianco FJ, Martinez-Salamanca JI. Focalyx Dx, Bx, Tx et Apps: A novel contemporary fusion paradigm for the management of prostate cancer. Arch Esp Urol. 2016 Jul;69(6):353-63. PMID 27416639
- [Background] Linares-Espinos E, Carneiro A, Martinez-Salamanca JI, Bianco F, Castro-Alfaro A, Cathelineau X, Valerio M, Sanchez-Salas R. New technologies and techniques for prostate cancer focal therapy. Minerva Urol Nefrol. 2018 Jun;70(3):252-263. doi: 10.23736/S0393-2249.18.03094-1. Epub 2018 Apr 16. PMID 29664243
- [Background] Gross MD, Sedrakyan A, Bianco FJ, Carroll PR, Daskivich TJ, Eggener SE, Ehdaie B, Fisher B, Gorin MA, Hunt B, Jiang H, Klein EA, Marinac-Dabic D, Montgomery JS, Polascik TJ, Priester AM, Rastinehad AR, Viviano CJ, Wysock JS, Hu JC. SPARED Collaboration: Patient Selection for Partial Gland Ablation in Men with Localized Prostate Cancer. J Urol. 2019 Nov;202(5):952-958. doi: 10.1097/JU.0000000000000357. Epub 2019 Oct 9. PMID 31144591
- [Background] Reis LO, Andrade DL, Bianco FJ Jr. Super active surveillance for low-risk prostate cancer | Opinion: Yes. Int Braz J Urol. 2019 Mar-Apr;45(2):210-214. doi: 10.1590/S1677-5538.IBJU.2019.02.02. No abstract available. PMID 31021584
- [Background] Ahdoot M, Lebastchi AH, Turkbey B, Wood B, Pinto PA. Contemporary treatments in prostate cancer focal therapy. Curr Opin Oncol. 2019 May;31(3):200-206. doi: 10.1097/CCO.0000000000000515. PMID 30865133
- [Background] Lodeizen O, de Bruin M, Eggener S, Crouzet S, Ghai S, Varkarakis I, Katz A, Dominguez-Escrig JL, Pahernik S, de Reijke T, de la Rosette J. Ablation energies for focal treatment of prostate cancer. World J Urol. 2019 Mar;37(3):409-418. doi: 10.1007/s00345-018-2364-x. Epub 2018 Jun 25. PMID 29943219
- [Background] Lindner U, Lawrentschuk N, Trachtenberg J. Focal laser ablation for localized prostate cancer. J Endourol. 2010 May;24(5):791-7. doi: 10.1089/end.2009.0440. PMID 20477544
- [Background] Chao B, Llukani E, Lepor H. Two-year Outcomes Following Focal Laser Ablation of Localized Prostate Cancer. Eur Urol Oncol. 2018 Jun;1(2):129-133. doi: 10.1016/j.euo.2018.03.011. Epub 2018 May 15. PMID 31100236
- [Background] Oto A, Sethi I, Karczmar G, McNichols R, Ivancevic MK, Stadler WM, Watson S, Eggener S. MR imaging-guided focal laser ablation for prostate cancer: phase I trial. Radiology. 2013 Jun;267(3):932-40. doi: 10.1148/radiol.13121652. Epub 2013 Feb 25. PMID 23440319